CLINICAL TRIAL: NCT00657995
Title: Continuous Postoperative Blood Glucose Monitoring and Control by an Artificial Pancreas in Patients Undergoing Pancreatic Resection: A Prospective Randomized Clinical Trial
Brief Title: Tight Glycemic Control by Artificial Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kochi University (Other)
Responsible Party: Kochi Medical School/Department of Surgery, Kochi University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGC-AP-01
Record Dates: First submitted 2008-04-04; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Pancreatic Neoplasm
Keywords: pancreatogenic; diabetes; artificial; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Diabetes Mellitus | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental): Thirty patients who underwent pancreatic resection for pancreatic neoplasm were prospectively randomized. Perioperative blood glucose levels were continuously monitored using an artificial endocrine pancreas (STG-22). Glucose levels were controlled using either the sliding scale method or the artificial pancreas.
  Interventions: Device: Artificial Pancreas (STG-22)

INTERVENTIONS:
Device: Artificial Pancreas (STG-22) — safe tool
  Other Names: STG-22; NIKKISO Corporation, Japan

SUMMARY:
This study evaluated a closed-loop system providing continuous monitoring and strict control of perioperative blood glucose following pancreatic resection.

DETAILED DESCRIPTION:
This study recruited 32 patients undergoing elective pancreatic resection for pancreatic disease.

ELIGIBILITY:
Inclusion Criteria:

* This study recruited 32 patients undergoing elective pancreatic resection for pancreatic disease.

Exclusion Criteria:

* weight loss greater than 10% during the previous 6 months
* signs of distant metastasis
* respiratory, renal,or heart disease
* Patients provided written informed consent prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
the incidence of severe hypoglycemia (< 40 mg/dl) during the intensive care period following pancreatic resection in patients monitored using the artificial pancreas | the first postoperative 18 hours in the surgical intensive care unit

SECONDARY OUTCOMES:
the total amount of insulin required for glycemic control after pancreatic resection | the first postoperative 18 hours in the surgical intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Takehiro Okabayashi, MD, Study Director — Kochi Medical School, Kochi University
Locations (1):
- Kochi Medical School, Kochi University, Nankoku, Kohasu-Okocho, Japan